CLINICAL TRIAL: NCT05921240
Title: Unmet Needs, Barriers and Facilitators to Vision Services for Children and Adolescents With Special Vision Care Needs: A Mixed-Model Design Study
Brief Title: Unmet Needs, Barriers and Facilitators to Vision Services for Children and Adolescents With Special Vision
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202305123RIND
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study, no intervention — no intervention

SUMMARY:
Children and adolescents with special needs, compared to those with general development, have a much higher incidence of visual impairments (10.5% vs. 0.16%). This project will focus on "children and adolescents with special visual care needs", comprehensively exploring their unmet needs in ophthalmology and visual care, as well as the obstacles and facilitators they may encounter in the process of seeking ophthalmic services.

The purposes of this study will investigate the current needs of children and adolescents with special visual care needs in ophthalmology and visual medical services, and the obstacles and potential facilitators encountered by children and adolescents with special visual care needs in the process of obtaining ophthalmology and visual medical services.

DETAILED DESCRIPTION:
The research will center on children and adolescents with special visual needs and explore the research questions from various stakeholders' perspectives, including parents, special education teachers and experts, healthcare professionals, workers from related NGOs and government units. A mixed-methods research approach will be used to gather both quantitative and qualitative data. After data analysis, a comparison and interpretation between the two results will be conducted to obtain the final research outcomes.

1. Quantitative research: Two-part questionnaire. The first part collects background information, and the second part is a "Needs and Difficulties Survey", framed by Levesque et al.'s conceptual framework of access to healthcare.
2. Qualitative research: The first part consists of semi-structured in-depth interviews, and the second part uses the focus group method. Both parts will use a common interview guideline and the International Classification of Functioning, Disability and Health, Child & Youth Version (ICF-CY) as the theoretical framework.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and fill out questionnaires in Chinese
2. Able to conduct interviews in Chinese

Exclusion Criteria:

1. The special needs children or adolescents they have taught do not have specific visual needs, hence they cannot provide relevant information.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents, educators, and profession with experience in children and adolescents with special needs in vision
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
qualitative data analysis | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Occupational Therapy, College of Medicine, Nation, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No